CLINICAL TRIAL: NCT06552585
Title: Effect of Two Preventive Exercise Programs for Swimmer's Shoulder on the Torque of Shoulder Rotator Muscles in Competitive Swimmers: a Randomized Controlled Trial
Brief Title: Effect of Two Preventive Exercise Programs for Swimmer's Shoulder on the Torque of Shoulder Rotator Muscles in Competitive Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Allied Health Sciences of Porto (ESTSP) - Polytechnic Institute of Porto (IPP) (Other)
Collaborators: University of Coimbra (Other); Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Nuno Tavares, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SchoolAHSP
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Pain; Injury;Sports; Sports Physical Therapy
Keywords: Swimmer's shoulder; Elastic band program; Weight program; Shoulder rotators; Injury prevention; Swimming
MeSH Terms: conditions — Shoulder Pain; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Care provider and participants blinded, parallel, randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: The physiotherapist who carried out the swimmer's interventions was external to the study. The participants were unaware of the existence of other sample groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight program group (Experimental)
  Interventions: Other: 12-weeks weight prevention program
- Elastic band program group (Experimental)
  Interventions: Other: 12-weeks elastic band prevention program
- Control (Sham Comparator)
  Interventions: Other: sham intervention

INTERVENTIONS:
Other: 12-weeks weight prevention program — Twice a week, over 12-weeks, the weight program group carried out a strength program with the 5 open kinetic chain exercises most often reported in the literature to prevent swimmer's shoulder - internal rotation at 90°, external rotation at 90°, scapular punches, T's, and Y's - with two weights Domyos with 1, 2, 3, 4, or 5 kg.The load used to perform the programs with weights were previously assessed and adjusted for each swimmer, corresponding to 75% of one repetition maximum. After 6 weeks of program execution, each swimmer carried out another one repetition maximum test assessment, to verify the possibility of a load instrument progression.
  Arms: Weight program group
Other: 12-weeks elastic band prevention program — Twice a week, over 12-weeks, the elastic band program group carried out a strength program with the 5 open kinetic chain exercises most often reported in the literature to prevent swimmer's shoulder - internal rotation at 90°, external rotation at 90°, scapular punches, T's, and Y's - with an elastic band Bodytone Power Band with 10, 15, 20, 25, or 30 kg weights Domyos.The load used to perform the programs with weights were previously assessed and adjusted for each swimmer, corresponding to 75% of one repetition maximum. After 6 weeks of program execution, each swimmer carried out another one repetition maximum test assessment, to verify the possibility of a load instrument progression.
  Arms: Elastic band program group
Other: sham intervention — The control group performed a sham intervention, twice a week, for 12-weeks. This intervention consisted of 2 sets of 10 repetitions of 5 shoulder mobility exercises, without preventive aim, normally carried out in warm-up before training: shoulder maximum flexion and extension, horizontal abduction and adduction starting from 90º of shoulder abduction, maximum internal/external rotation starting from 90º of shoulder abduction, circumduction of the shoulder in a clockwise direction and circumduction of the shoulder in a counterclockwise direction. There was no progression after 6-weeks of this sham intervention. The coach of the respective team checked the execution of the exercises, but there was no individualized monitoring with a regular exercise technique correction by a physiotherapist.
  Arms: Control

SUMMARY:
The purpose of this study was to verify the effectiveness of two 12-week preventive exercise programs for swimmer's shoulder with monitoring and progression over time, on the peak torque and respective conventional concentric ratio and functional ratio. One of these programs was performed with weights and the other with an elastic band. This study hypothesized that the two preventive exercise programs minimize shoulder rotators imbalanced during the swimming season. The study design is a care provider and participants blinded, parallel, randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Competitve swimmer in the current season.
* Aged between 16-35 years old.
* Have a minimum of 5 years of experience in national competitions.
* Performed a minimum of 8 hours of weekly swimming training.

Exclusion Criteria:

* Subjects who had performed at least 6 weeks of treatment such as physical therapy, injections, and medication.
* Clinical situations such as a history of significant shoulder pain in the last 6 months, a history of traumatic shoulder injuries such as fractures, subluxations, cervical or thoracic conditions, previous shoulder surgeries, shoulder range of motion deficits, or neurological injuries.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Peak torque | 12 weeks
  The concentric and eccentric peak torque of internal and external rotators of the dominant and non-dominant shoulders at 60°/s, 120°/s and 180°/s, evaluated through an isokinetic dynamometer Biodex System 3 (Biodex Medical Systems, New York).

SECONDARY OUTCOMES:
Conventional concentric external/internal shoulder rotators ratio | 12 weeks
  The quotient between peak torque values of the concentric external and internal rotators of the shoulder multiplied by 100.
Functional eccentric external/concentric internal shoulder rotators ratio | 12 weeks
  The quotient between peak torque values of the eccentric external rotators of the shoulder and concentric internal rotators of the shoulder multiplied by 100.
Time to peak torque | 12 weeks
  The time between the beginning of the torque caption and the peak torque previously described.

CONTACTS AND LOCATIONS:
Overall Officials: Maria António Castro, PhD, Study Director — Instituto Politécnico de Leiria
Locations (1):
- Instituto Politécnico de Coimbra - RoboCorp, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavares N, Vilas-Boas JP, Castro MA. Effect of Preventive Exercise Programs for Swimmer's Shoulder Injury on Rotator Cuff Torque and Balance in Competitive Swimmers: A Randomized Controlled Trial. Healthcare (Basel). 2025 Mar 1;13(5):538. doi: 10.3390/healthcare13050538. PMID 40077099

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT06552585/Prot_SAP_000.pdf